CLINICAL TRIAL: NCT04188821
Title: Reduction of Seroma and Improvement of Quality of Life After Early Drain Removal in Immediate Breast Reconstruction With Tissue Expander. Preliminary Report of a Randomized Controlled Study
Brief Title: Reduction of Seroma and Improvement of QoL in Breast Reconstruction With Tissue Expander
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Lembo Fedele, Principal Investigator, University of Foggia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01/2019
Record Dates: First submitted 2019-11-28; First posted 2019-12-06 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Safety Issues; Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- output based group (Active Comparator): Investigators remove the drains when the suction drain flow was less than 30 ml/day for at least 2 days with no further signs of infection, fluid collection or impaired wound healing
  Interventions: Procedure: breast drain removal
- early-removal group (Experimental): Investigators remove the drains at hospital discharge, 3-4 days after surgery, regardless of the output at that time
  Interventions: Procedure: breast drain removal

INTERVENTIONS:
Procedure: breast drain removal — Investigators remove the drains when the suction drain flow was less than 30 ml/day for at least 2 days or at discharge, with no further signs of infection, fluid collection or impaired wound healing ("complicated", see below). Ultimately, we removed drains 3 weeks postoperatively (21 days post op) even if the flow was higher than 30 ml/day. However, leakage or severe patient discomfort led to immediate drain removal at any time during postoperative care.

SUMMARY:
The experimental hypothesis of this randomized controlled study was to demonstrate that early drain removal in patients who underwent immediate breast reconstruction with tissue expander is a safety procedure to improving clinical outcomes and quality of life (QoL). The mechanism of action underlying the proposed approach was intuitive. The early drain removal allows to: 1) avoid continuous seroma development caused by active suction of drain (stopping the circle "drain itself may perpetuate the drainage" with vacuum mechanism); 2) reduce the risks connected to "foreign body reaction" as tissue inflammation and infection; 3) improve QoL reducing pain, length of hospital stay and limitations of daily activities.

ELIGIBILITY:
Inclusion Criteria:

* SNS (skin nipple sparing) or SS (skin sparing) mastectomy for breast cancer and immediate positioning of breast expander (without mesh) with placement of suction drain, regardless of TNM classification

Exclusion Criteria:

* skin reducing mastectomy, reconstruction with flap, direct to implant reconstruction (with or without mesh or ADM) and axillary dissection

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
total fluid volume (ml) | 21 days
  sum of drain volumes and volume of seroma aspirations if needed
days with drainage | 21 days
days of seroma formation | 21 days
  period that drain or seroma aspiration is needed in days after surgery
time until wound healing (days) | 21 days
infection (yes or not) | 21 days
  defined as the appearance of local signs/symptoms as erythema, edema, induration, increased pain, and a change in drainage to a purulent nature and fever, confirmed by swabs
complicated wound healing (yes or not) | 21 days
  unclosed wound 3 weeks postoperatively

SECONDARY OUTCOMES:
pain (using Visual Analogic Score scale to measure intensity) | 21 days
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain." (10)
disturbance in quality of sleep (yes or not) | 21 days
limitation in personal care, daily activities and social life (yes or not) | 21 days
disturbance in mobility (yes or not) | 21 days
  mobility as walking, running, driving

IPD SHARING:
Plan to Share IPD: Undecided